CLINICAL TRIAL: NCT03345719
Title: The Translational Research Image-Guided Operating Room (TRIGORA): Intraoperative 3D Imaging for Head & Neck Surgical Patients
Acronym: TRIGORA
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 12-5315
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 3D Cone-Beam Imaging

SUMMARY:
Head and neck cancer surgery presents the challenge of tumour resection in close proximity to critical structures such as the carotid arteries and optic nerves. The need for precise localization within complex 3D anatomy has motivated the development of image-guidance systems that account for tissue deformation and excision through the use of intraoperative cone-beam CT (CBCT). A prototype mobile C-arm for intraoperative flat-panel CBCT has been developed at UHN in collaboration with Siemens Healthcare to provide low-dose 3D images with sub-mm spatial resolution and soft-tissue visibility. Extensive investigation in pre-clinical/clinical H&N, otology, orthopaedic, lung, and spine surgery has demonstrated the benefit of intraoperative CBCT for improved target ablation, localization accuracy, and critical structure avoidance.

Prospective clinical trial in CBCT-guided H&N surgery will be conducted to evaluate the Zeego robotic platform for CBCT. Patient accrual will span a wide range of surgical procedures in otolaryngology, including cancer resection and anatomical reconstruction in the mandible, maxilla, sinuses, skull base, and temporal bone. The effect of intraoperative imaging and surgical guidance on logistical considerations of time, workflow, and compatibility with the OR environment will be evaluated through the use of in-room audio/video recordings, human factors engineering methods, and expert feedback questionnaires obtained from the surgeons, nurses, and anesthetists involved in each case. This clinical investigation will help to further define indications for CBCT-guided H&N surgery, and serve to enable the development of surgical task-specific imaging protocols.

DETAILED DESCRIPTION:
For each patient enrolled in this study, the following administrative information will be compiled and maintained by the Principal Investigator at Princess Margaret Hospital:

Consent Form: The signed consent form. (Note that the Consent Form is the only information collected in this study that is not anonymous. All subsequent information is identified by an arbitrary Code # that can not be directly or indirectly traced back to the individual patient.) Clinical Summary: A brief summary provided by the Clinical Co-Investigator and/or Surgical Fellow regarding the patient's illness and prescribed surgical treatment plan. The Clinical Summary is anonymous with respect to patient identity and will be identified by an arbitrary Code #. The Summary will include age, weight, height, sex, diagnosis, stage, habits (viz., smoking and alcohol consumption), results of physical examination, and relevant medical history (e.g., prior surgery). This will also include medical history related to suitability for IV contrast (see the form included with the protocol).

Procedure Log: A summary log of the surgical procedure and imaging studies, when and where they were carried out, and relevant notes regarding the surgical and imaging procedures therein e.g., success or failure of the treatment plan or imaging system, etc. The Procedure Log is also anonymous and identified by an arbitrary Code #.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients with tumors or other masses in the following sites, nasal cavity, sinuses, nasopharynx, parapharyngeal space, deep parotid salivary glands, oral cavity, oropharynx, and skull base. Cases considered in this study will include lesions in one or several of these sites.

The patients are intended to undergo surgical treatment for their disease. The patients should have a complete and detailed medical record. Subjects must be at least 18 years of age. Subjects must sign and be given a copy of the written Informed Consent Form.

Exclusion Criteria:

* Patients with unresectable lesions, where surgery is not the treatment of choice.

Patients who are not able to consent by themselves or grasp the implication of the study.

Subjects participating in any other clinical trial during the time of this clinical investigation and that may have an impact on this evaluation.

Subjects may be excluded from this study at the discretion of a Clinical Co-Investigator, if they are enrolled in other studies that will result in combined radiation exposure exceeding standard of care.

Subjects who are pregnant, lactating, or planning to become pregnant during the period of the evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery to the head and neck and deemed eligible for this study by the investigators.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2012-10-04 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of 3D cone-beam imaging | intraoperative
  Evaluate the performance of 3D cone-beam imaging in the operating room

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada